CLINICAL TRIAL: NCT01814267
Title: Medico-economical Assessment of Telemedicine During Chronic Diabetes-related Foot Wound Management
Acronym: AIRPEDIA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurCIC, Pr Pierre-Yves BENHAMOU, University Hospital, Grenoble, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 12 07
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Diabetes; Diabetic Foot Ulcer
Keywords: innovative care; telemedicine; cost effectiveness; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Telemedicine; Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemedicine (Experimental): care and follow-up through telemedicine.
  Interventions: Other: telemedicine
- Conventional care (Active Comparator): care and follow-up through iterative diabetes physician consultations (conventional care and follow-up)
  Interventions: Other: conventional

INTERVENTIONS:
Other: telemedicine — Intervention group: care and follow-up through telemedicine (e-consultations)
  * 1 hospital consultation at inclusion time, week 0
  * then every 15 days, after the transmission of medical data and photos via internet by the nurse, telemedicine e-consultations until the wound has healed (week 2,week 4, week 6, week 8, week 10, week 12, week 14, week 16, week 18, week 20, week 22, week 24 : end point study), i.e. 12 e-consultations over a 6-month period.
  * 1 hospital consultation to validate that the wound is well-healed
  Arms: Telemedicine
Other: conventional — conventional group: iterative diabetes physicians consultations at hospital
  * 1 consultation at inclusion time, week 0
  * 1 consultation 2 weeks after inclusion, week 2
  * 1 consultation per month until the wound has healed (week 4, week 8, week 12, week 16, week 20, week 24: end-point study), i.e. 6 consultations over a 6-month period
  * 1 consultation to validate that the wound is well-healed
  Arms: Conventional care

SUMMARY:
The aim of the study is to assess the cost-effectiveness of telemedicine in the care of chronic diabetic foot ulcers.

Patients will be randomized into 2 groups: 1/conventional care group with iterative visits to diabetes specialist or 2/innovative care (telemedicine group).

the health insurance system perspective is adopted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or 2 diabetes, at least 18 years old
* Patient with a diabetic foot wound :

  * Acute or chronic (evolving for at least 30 days)
  * size ≤ to 3 cm²
  * Level I, II or III, stage A or B, excluding stages C and D from the University of Texas Wound Classification Systems
* Person affiliated to French Health insurance or equivalent
* Person having signed freely the consent form after receiving sufficient information
* Treatment compliance and 6 months follow-up feasible

Exclusion Criteria:

* Patient with a ischemic wound: Ankle-Brachial Index (ABI) <0.9 or Transcutaneous oxygen pressure (TcpO2) < 30 mmHg (stage C and D from the University of Texas Wound Classification Systems)
* Patient with emergency hospitalization indication whatever the reasons.
* Person deprived of liberty by a legal or administrative decision, patients in emergency and people hospitalised without consent and who are not protected by law.
* Pregnant or breastfeeding women
* Patient currently participating in another telemedicine research protocol (such as : Study on the impact of Telemedicine on the management of patients with type 1 diabetes (TELEDIAB-3))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Assess the incremental cost-effectiveness ratio from the french health system perspective | 6 months
  It is elaborated from:
  1. Main cost criteria: transport, outpatient costs (home nursing care, physicians consultations...), loss of productivity (absence from work)
  2. Main clinical effectiveness criterion: wound healing time.

SECONDARY OUTCOMES:
Assess the Impact of telemedicine care from the hospital perspective | 6 months
  The incremental cost-effectiveness ratio is calculated from the hospital perspective:
  1. Main cost criteria will be collected according to the micro-costing method: costs of innovative medical device (implementation and maintenance of telemedicine platform), telemedicine physician consultations, standard consumables, cost of care rooms and cost of medical and paramedical staff and, standard consumables for wound treatment.
     Costs will not include structural costs
  2. Main clinical effectiveness criterion: wound healing time
Assess acceptability of telemedicine care (compliance and satisfaction) for patients and nurses. | 6 months
  Acceptability questionnaire for nurse including use or misuse of telemedicine. Acceptability questionnaire for patient.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves BENHAMOU, MD PHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Hazenberg CE, Bus SA, Kottink AI, Bouwmans CA, Schonbach-Spraul AM, van Baal SG. Telemedical home-monitoring of diabetic foot disease using photographic foot imaging--a feasibility study. J Telemed Telecare. 2012 Jan;18(1):32-6. doi: 10.1258/jtt.2011.110504. Epub 2011 Nov 8. PMID 22067285
- [Background] Foltynski P, Ladyzynski P, Migalska-Musial K, Sabalinska S, Ciechanowska A, Wojcicki J. A new imaging and data transmitting device for telemonitoring of diabetic foot syndrome patients. Diabetes Technol Ther. 2011 Aug;13(8):861-7. doi: 10.1089/dia.2011.0004. Epub 2011 May 13. PMID 21568750
- [Background] Bowling FL, King L, Paterson JA, Hu J, Lipsky BA, Matthews DR, Boulton AJ. Remote assessment of diabetic foot ulcers using a novel wound imaging system. Wound Repair Regen. 2011 Jan-Feb;19(1):25-30. doi: 10.1111/j.1524-475X.2010.00645.x. Epub 2010 Dec 6. PMID 21134035
- [Background] Larsen SB, Clemensen J, Ejskjaer N. A feasibility study of UMTS mobile phones for supporting nurses doing home visits to patients with diabetic foot ulcers. J Telemed Telecare. 2006;12(7):358-62. doi: 10.1258/135763306778682323. PMID 17059653
- [Background] Wilbright WA, Birke JA, Patout CA, Varnado M, Horswell R. The use of telemedicine in the management of diabetes-related foot ulceration: a pilot study. Adv Skin Wound Care. 2004 Jun;17(5 Pt 1):232-8. doi: 10.1097/00129334-200406000-00012. PMID 15192491
- [Result] Muller M, David-Tchouda S, Margier J, Oreglia M, Benhamou PY. Comment on Rasmussen et al. A Randomized Controlled Trial Comparing Telemedical and Standard Outpatient Monitoring of Diabetic Foot Ulcers. Diabetes Care 2015;38:1723-1729. Diabetes Care. 2016 Jan;39(1):e9-10. doi: 10.2337/dc15-1659. No abstract available. PMID 26696670